CLINICAL TRIAL: NCT04608773
Title: Evaluation of Two Mouth Sprays for Post-irradiation Xerostomia in Head and Neck Cancer Survivors: a Randomized, Double-blind Clinical Trial
Brief Title: Blinded Dry Mouth Spray Crossover Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonas Johnson (Other)
Collaborators: TJA Health, LLC (Industry)
Responsible Party: Sponsor-Investigator, Jonas Johnson, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: STUDY20090008
Record Dates: First submitted 2020-10-18; First posted 2020-10-29 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Xerostomia; Head and Neck Cancer; Xerostomia Following Radiotherapy
Keywords: Mouth Spray
MeSH Terms: conditions — Xerostomia; Head and Neck Neoplasms | interventions — Xylitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both subjects and clinicians will be blinded to Mouth Spray A and Mouth Spray B.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Biotene Spray, followed by Refresh Spray (Other): The Biotene Spray followed by Refresh Spray Arm will be asked to complete a 2 week trial using Biotene Spray first, then will be asked to complete a 2 week trial using Refresh Spray second. (after the appropriate 1 week washout periods have been completed)
  Interventions: Other: Remineralizing Extreme Dry Mouth Spray with Xylitol; Device: Alcohol-Free Moisturizing Dry Mouth Spray
- Refresh Spray, followed by Biotene Spray (Other): The Refresh Spray, followed by Biotene Spray Arm will be asked to complete a 2 week trial using Refresh Spray first, then will be asked to complete a 2 week trial using Biotene Spray second. (after the appropriate 1 week washout periods have been completed)
  Interventions: Other: Remineralizing Extreme Dry Mouth Spray with Xylitol; Device: Alcohol-Free Moisturizing Dry Mouth Spray

INTERVENTIONS:
Other: Remineralizing Extreme Dry Mouth Spray with Xylitol — oral hydrating spray
  Other Names: Refresh Oral Hydrating Spray
Device: Alcohol-Free Moisturizing Dry Mouth Spray — oral hydrating spray
  Other Names: Biotene

SUMMARY:
To identify the effectiveness of two mouth sprays at relieving symptoms of xerostomia in patients who have received radiation for carcinoma of the head and neck.

To assess patient quality of life and mouth acidity following use of two mouth sprays meant to relieve symptoms of xerostomia in patients who have received radiation for carcinoma of the head and neck.

DETAILED DESCRIPTION:
Investigators have observed that patients at the University of Pittsburgh Medical Center Head and Neck Survivorship clinic with symptoms of radiation-induced xerostomia expressed verbal preference for Biotene and Refresh mouth sprays (spray form of mouthwash) compared to other oral products such as gel, toothpaste, and chewing gum. Investigators have designed this study to specifically assess the effectiveness of mouth sprays on xerostomia in patients who have completed radiation for head and neck carcinoma. While there have been clinical trials to evaluate the effectiveness of Biotene oral products for xerostomia, Refresh mouthwash/mouth spray is a newer oral rinse formula that has not undergone any randomized controlled trials to evaluate its efficacy compared to other agents of its kind. The investigators have put forward this randomized controlled trial to compare the efficacy of both sprays to each other and to water. Biotene spray is cleared by the FDA as a medical device product. Currently, Refresh mouth spray falls under the FD&C Act.

There is preliminary data on the effectiveness of Biotene mouthwash for xerostomia in patients who have had radiation of the head and neck. A phase II study of Biotene products (mouthwash, chewing gum, and toothpaste) were effective at improving many symptoms of post-irradiation xerostomia. Numerous other studies have shown that mouthwash and topical dry mouth products improve xerostomia symptoms.

Xerostomia, or mouth dryness, is a frequent side effect of head and neck cancer radiation therapy, as the salivary glands are often damaged during therapy. Radiation therapy can be successful in treating cancer, but post-irradiation xerostomia can cause oral discomfort as well as issues with eating, speech, and oral hygiene, leading to significantly decreased quality of life. While treatment of xerostomia has limited benefit, various mouthwashes have led to major symptomatic improvement in some patients. This study will add to existing literature by commenting on efficacy of a popular and established mouth spray used for xerostomia as well as a new mouth spray that has not been compared to existing formulas. A double-blinded randomized controlled trial evaluating these mouth sprays will add information about value of both formulas for head and neck carcinoma survivors with radiation-induced xerostomia.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-proven oral cavity, oropharynx, larynx, and hypopharynx carcinoma
* who received primary radiation with curative intent (>50 Gray in 20 fractions)
* radiation treatment completed greater than 6 months ago
* who endorse xerostomia

Exclusion Criteria:

* evidence of metastasis or recurrent disease
* Current use of pilocarpine, antidepressants, anticholinergic drugs, or any other medication that has an effect on salivation
* those who have documented medical conditions associated with xerostomia such as Sjogren's Syndrome
* those who use oral inhalants for the treatment of respiratory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonas T Johnson, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epstein JB, Emerton S, Le ND, Stevenson-Moore P. A double-blind crossover trial of Oral Balance gel and Biotene toothpaste versus placebo in patients with xerostomia following radiation therapy. Oral Oncol. 1999 Mar;35(2):132-7. doi: 10.1016/s1368-8375(98)00109-2. PMID 10435146
- [Background] Warde P, Kroll B, O'Sullivan B, Aslanidis J, Tew-George E, Waldron J, Maxymiw W, Liu FF, Payne D, Cummings B. A phase II study of Biotene in the treatment of postradiation xerostomia in patients with head and neck cancer. Support Care Cancer. 2000 May;8(3):203-8. doi: 10.1007/s005200050286. PMID 10789961
- [Background] Eisbruch A, Rhodus N, Rosenthal D, Murphy B, Rasch C, Sonis S, Scarantino C, Brizel D. How should we measure and report radiotherapy-induced xerostomia? Semin Radiat Oncol. 2003 Jul;13(3):226-34. doi: 10.1016/S1053-4296(03)00033-X. PMID 12903012

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1824 patients were screened for eligibility at UPMC's Head and Neck Cancer Survivorship Clinic between January 2021 and September 2022.
Pre-assignment Details: 468 patients were found eligible, 339 declined to participate and 129 were enrolled.
Period: First Wash Out (1 Week)
Arm/Group | Biotene Spray, Followed by Refresh Spray | Refresh Spray, Followed by Biotene Spray
Started | 69 | 60
Completed | 57 | 54
Not Completed | 12 | 6
Not completed — Withdrawal by Subject | 12 | 6
Period: First Intervention (2 Weeks)
Arm/Group | Biotene Spray, Followed by Refresh Spray | Refresh Spray, Followed by Biotene Spray
Started | 57 | 54
Completed | 53 | 50
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 3 | 1
Not completed — mild adverse effects | 1 | 3
Period: Second Wash Out (1 Week)
Arm/Group | Biotene Spray, Followed by Refresh Spray | Refresh Spray, Followed by Biotene Spray
Started | 53 | 50
Completed | 53 | 50
Not Completed | 0 | 0
Period: Second Intervention (2 Week)
Arm/Group | Biotene Spray, Followed by Refresh Spray | Refresh Spray, Followed by Biotene Spray
Started | 53 | 50
Completed | 51 | 45
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 2 | 4
Not completed — mild adverse effect | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biotene Spray, Followed by Refresh Spray | Refresh Spray, Followed by Biotene Spray | Total
Number analyzed (Participants) | 69 | 60 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 31 | 66
  >=65 years | 34 | 29 | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 55 | 48 | 103
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only participants who completed the protocol were included in the analysis.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 4 | 5
    White | 68 | 56 | 124
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 69 | 60 | 129
Drymouth baseline [Mean (Standard Deviation); unit: units on a scale] — Patients responded to electronic survey; the questionnaire included continuous variables derived from the 100mm visual analog scale (VAS). "During the last three days, overall, your mouth or tongue was: 'Very Dry' = 0 10 20 30 40 50 60 70 80 90 100 = 'Not at All Dry"
  units on a scale | 44.0 (20.6) | 39.2 (21.8) | 42.4 (21.0)

OUTCOME MEASURES:

1. Primary Outcome: Oral Dryness
Description: at the end of each study period an online questionnaire was administered. The questionnaire included continuous variables derived from the 100mm visual analog scale (VAS); documented via questionnaire completion by participants administered via Qualtrics.
  Dryness was measured on a 0-100 point scale "During the last three days, overall, your mouth or tongue was: 'Very Dry' = 0 10 20 30 40 50 60 70 80 90 100 = 'Not at All Dry"
Time Frame: 2 week trial period
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Biotene Spray: Participants who received Biotene in either the first or last two week trial period of the study.
- Refresh Spray: Participants who received Refresh spray in either the first or second two week period of the study.
Arm/Group | Biotene Spray | Refresh Spray
Number analyzed (Participants) | 96 | 96
units on a scale
  Oral dryness Dryness baseline | 45.5 (20.3) | 46.6 (22.7)
  Dryness 2 weeks | 52.76 (19.25) | 54.1 (21.6)
Statistical Analysis 1: Comparison: Biotene Spray vs Refresh Spray; Null hypothesis is that there was no difference in change of Dry mouth score between Refresh and Biotene. ANCOVA model was performed by regressing the difference in after-treatment measurement between Refresh and Biotene over the difference of baseline between Refresh and Biotene. The test was performed with a significance level of 0.05 (two- sided); Test type: Superiority; p < 0.501, ANCOVA

2. Secondary Outcome: Sleeping Difficulty Due to Oral Dryness
Description: sleeping difficulty due to oral dryness was documented via questionnaire completion by participants administered via Qualtrics. Sleeping difficulty will be measured on a 0-100 point scale
  "During the last three days, due to the dryness of your mouth and tongue, how difficult was it to sleep? Consider such factors as how difficult it was for you to go to sleep, the duration and quality of your sleep, and how often you woke up to drink or urinate. Very Difficult 0 10 20 30 40 50 60 70 80 90 100 Easy" (Higher score means better outcome)
Time Frame: 2 week trial
Population: Number of participants in analysis is less than overall number of participants due to missing responses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Biotene Spray: Participants who received Biotene spray either in the first or last 2 week trial period.
- Refresh Spray: Participants who received Refresh spray either in the first or second 2 week trial period.
Arm/Group | Biotene Spray | Refresh Spray
Number analyzed (Participants) | 96 | 96
units on a scale
  Sleep Baseline: number analyzed (Participants) | 90 | 90
  Sleep Baseline | 56.3 (27.0) | 61.9 (26.3)
  Sleep 2 weeks | 66.8 (23.0) | 64.8 (24.9)
Statistical Analysis 1: Comparison: Biotene Spray vs Refresh Spray; Test type: Superiority; p = .109, ANCOVA

3. Secondary Outcome: Speaking Difficulty Due to Oral Dryness
Description: Speaking difficulty due to oral dryness was documented via questionnaire completion by participants administered via Qualtrics. Speaking difficulty will be measured on a 0-100 point scale "During the last three days, due to the dryness of your mouth and tongue, how difficult was it to speak without drinking liquids? Very Difficult 0 10 20 30 40 50 60 70 80 90 100 Easy"
Time Frame: 2 week trial
Population: The number of participants in analysis are lower in this specific analysis due to missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Speaking Difficulty Score After Biotene Spray: Participants who received Biotene in either the first or last two week trial period of the study.
- Speaking Difficulty Score After Refresh Spray: Participants who received Refresh spray in either the first or second two week period of the study.
Arm/Group | Speaking Difficulty Score After Biotene Spray | Speaking Difficulty Score After Refresh Spray
Number analyzed (Participants) | 96 | 96
units on a scale
  speaking baseline: number analyzed (Participants) | 91 | 91
  speaking baseline | 60.8 (27.6) | 63.0 (26.6)
  speaking 2 weeks | 69.9 (22.2) | 66.8 (24.1)
Statistical Analysis 1: Comparison: Speaking Difficulty Score After Biotene Spray vs Speaking Difficulty Score After Refresh Spray; Test type: Superiority; p = .107, ANCOVA

4. Secondary Outcome: Taste Alteration/Impairment Due to Oral Dryness
Description: Alteration/impairment in sense of taste will be documented via questionnaire completion by participants administered via Qualtrics. Taste alteration/impairment will be measured on a 0-100 point scale "During the last three days, has your sense of taste been impaired or affected? Greatly Impaired/Affected 0 10 20 30 40 50 60 70 80 90 100 Not Impaired/Affected"
Time Frame: 2 week trial
Population: The number of participants in this analysis are lower than the overall population due to missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Biotene Spray Trial: Participants who received Biotene in either the first or last two week trial period of the study.
- Refresh Spray Trial: Participants who received Refresh spray in either the first or second two week trial period of the study.
Arm/Group | Biotene Spray Trial | Refresh Spray Trial
Number analyzed (Participants) | 96 | 96
units on a scale
  Taste baseline: number analyzed (Participants) | 91 | 91
  Taste baseline | 73.2 (29.0) | 71.5 (29.3)
  Taste 2 weeks | 78.1 (22.8) | 75.4 (27.0)
Statistical Analysis 1: Comparison: Biotene Spray Trial vs Refresh Spray Trial; Test type: Superiority; p = .489, ANCOVA

5. Secondary Outcome: Swallowing and Chewing Difficulty Due to Oral Dryness
Description: Swallowing and chewing difficulty due to oral dryness will be documented via questionnaire completion by participants administered via Qualtrics. Swallowing and chewing difficulty will be measured on a 0-100 point scale "During the last three days, overall, due to the dryness of your mouth and tongue, how difficult was it to chew and swallow food? Very Difficult 0 10 20 30 40 50 60 70 80 90 100 Easy"
Time Frame: 2 week trial
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biotene Spray Trial | Refresh Spray Trial
Number analyzed (Participants) | 96 | 96
units on a scale
  swallowing baseline | 53.7 (25.6) | 54.6 (24.4)
  swallowing 2 weeks | 62.7 (24.1) | 60.4 (23.4)
Statistical Analysis 1: Comparison: Biotene Spray Trial vs Refresh Spray Trial; Test type: Superiority; p = .213, ANCOVA

6. Secondary Outcome: Saliva PH
Description: PH Is a measure of acidity on a logarithmic scale range 0 (most acidic) to 14 (most basic) with a neutral PH of 7 as the desired outcome.
Time Frame: 2 week trial
Population: The number of participants in this analysis are lower than the overall population due to missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biotene Spray Trial | Refresh Spray Trial
Number analyzed (Participants) | 96 | 96
units on a scale
  PH baseline: number analyzed (Participants) | 91 | 91
  PH baseline | 5.3 (1.0) | 5.5 (1.1)
  PH 2 weeks | 5.4 (1.0) | 5.5 (1.1)
Statistical Analysis 1: Comparison: Biotene Spray Trial vs Refresh Spray Trial; Test type: Superiority; p = .486, ANCOVA

7. Secondary Outcome: Difficulty Wearing Dental Prostheses (if Applicable)
Description: Difficulty wearing dental prostheses (if applicable) will be documented via questionnaire completion by participants administered via Qualtrics. Dental prostheses wearing difficulty will be measured on a 0-100 point scale "If you normally wear dentures, due to the dryness of your mouth and tongue, how difficult was it to wear dentures during the last three days? (If you do not normally wear dentures or could not wear dentures for other reasons not associated with dry mouth, please check the box marked "Not applicable") Very Difficult 0 10 20 30 40 50 60 70 80 90 100 Easy Not Applicable
Time Frame: 6 weeks
Population: No participants in study with dental prosthesis, therefore data was not collected.
Groups:
- Difficulty Wearing Dental Prosthesis Score After Biotene Spray: Participants who received Biotene in either the first or last two week trial period of the study.
- Difficulty Wearing Dental Prosthesis Score After Refresh Spray: Participants who received Refresh spray in either the first or second two week period of the study.
Arm/Group | Difficulty Wearing Dental Prosthesis Score After Biotene Spray | Difficulty Wearing Dental Prosthesis Score After Refresh Spray
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Biotene Spray: Participants who received biotene spray in either the 1st or 2nd two week trial period
- Refresh Spray: Participants who received Refresh spray in either the 1st or 2nd two week trial period
Arm/Group | Biotene Spray | Refresh Spray
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/129
Serious Adverse Events (participants affected / at risk) | 0/129 | 0/129
Other Adverse Events (participants affected / at risk) | 0/129 | 5/129
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Biotene Spray (N=129) | Refresh Spray (N=129)
oral burning and swelling sensation (Skin and subcutaneous tissue disorders) | 0 | 5

LIMITATIONS AND CAVEATS:
There may be a degree of attrition bias, our modified intention-to-treat design, in which 13 patients had to be reassigned to group 1 from group 2, may have also added bias; we found no evidence of a sequence effect. The treatment effect of each spray was calculated in reference to use of water, which is known to improve oral dryness so the magnitude of the treatment effect may be underestimated, however, we would expect both products to be affected equally.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT04608773/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT04608773/ICF_001.pdf